CLINICAL TRIAL: NCT04511598
Title: Precision of 3 Dimensional Facial Analysis Using Bellus 3D Face Camera Pro Versus Planmeca ProMax 3D Proface: A Diagnostic Accuracy Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sally Faisal Mahmoud Fouad Abdallah, Masters Degree Student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: ORTH 7-1-2
Record Dates: First submitted 2020-08-09; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: 3 Dimensional Soft Tissue Facial Analysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bellus 3D Face Camera Pro (Experimental): Every single patient will be diagnosed using 3D imaging system "Bellus 3D Face Camera Pro" to be compared to the direct measurements obtained from direct anthropometry.
  Interventions: Device: "Bellus 3D Face Camera"; Device: "Planmeca ProMax 3D Proface"
- Planmeca ProMax 3D Proface (Experimental): Every single patient will be diagnosed using 3D imaging systems "Planmeca ProMax 3D Proface" to be compared to the direct measurements obtained from direct anthropometry.
  Interventions: Device: "Bellus 3D Face Camera"; Device: "Planmeca ProMax 3D Proface"

INTERVENTIONS:
Device: "Bellus 3D Face Camera" — The depth sensor uses infrared structured light scanning technology to capture depth and the camera on the phone or tablet to capture color texture of the face.
Device: "Planmeca ProMax 3D Proface" — The lasers scan the facial geometry and the digital cameras capture the color texture of the face.

SUMMARY:
Precision of 3 Dimensional Facial Analysis Using "Bellus 3D Face Camera Pro" Versus "Planmeca ProMax 3D Proface" is to be evaluated in comparison to direct anthropometry.

DETAILED DESCRIPTION:
The aim of this study will be the evaluation of the precision and reproducibility of standard anthropometric linear measurements made with two different three-dimensional imaging systems namely "Bellus 3D Face Camera Pro" and "Planmeca ProMax 3D ProFace system" and to compare them to physical linear measurements "Direct Anthropometry".

ELIGIBILITY:
Inclusion Criteria:

1. Age range from 18-35 years.
2. Normal balanced facial proportions.

Exclusion Criteria:

1. Craniofacial anomalies.
2. Obvious skeletal shifts.
3. Patients with incompetent lips.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Precision | 1 Month
  Evaluation of the precision of standard anthropometric linear measurements made with two different three-dimensional imaging systems namely Bellus 3D Face Camera Pro and Planmeca ProMax 3D ProFace system and to compare them to physical linear measurements.

SECONDARY OUTCOMES:
Reproducibility | 1 Month
  Evaluation of the reproducibility of standard anthropometric linear measurements made with two different three-dimensional imaging systems namely Bellus 3D Face Camera Pro and Planmeca ProMax 3D ProFace system and to compare them to physical linear measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo, Giza Governorate, Egypt